CLINICAL TRIAL: NCT03875326
Title: Testing High Definition Transcranial Direct Current Stimulation (HD-tDCS) as Treatment of Mild Cognitive Impairment
Brief Title: Stimulation to Improve Memory
Acronym: STIM
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Michigan (Other)
Collaborators: National Institute on Aging (NIA) (NIH)
Responsible Party: Principal Investigator, Benjamin Hampstead, PhD, Stanley Berent, Ph.D., Collegiate Professor of Psychology, University of Michigan
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: HUM00146180; 1R01AG058724 (NIH)
Record Dates: First submitted 2019-03-11; First posted 2019-03-14 (Actual); Last update posted 2025-10-20 (Actual); Status verified 2025-10

CONDITIONS: Mild Cognitive Impairment; Dementia of Alzheimer Type
Keywords: Dementia; Memory; Cognitive Rehabilitation; PET scan; fMRI; Brain Stimulation
MeSH Terms: conditions — Cognitive Dysfunction; Dementia

STUDY DESIGN:
Intervention Model Description: Eligible participants will be randomized 1:1:1:1 to receive either sham, 1mA, 2mA, or 3mA HD-tDCS for at least 5 sessions and up to 30 sessions using a blocked randomization design.
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (4):
- Sham Stimulation (Sham Comparator): Sham (placebo) dose of HD-tDCS treatment for 30 minutes, for between 5-30 sessions.
  Interventions: Device: Sham
- 1 mA Dosage Stimulation (Experimental): 1 milliAmp dose of HD-tDCS treatment for 30 minutes, for between 5-30 sessions.
  Interventions: Device: 1 mA HD-tDCS
- 2 mA Dosage Stimulation (Experimental): 2 milliAmp dose of HD-tDCS treatment for 30 minutes, for between 5-30 sessions.
  Interventions: Device: 2 mA HD-tDCS
- 3 mA Dosage Stimulation (Experimental): 3 milliAmp dose of HD-tDCS treatment for 30 minutes, for between 5-30 sessions.
  Interventions: Device: 3 mA HD-tDCS

INTERVENTIONS:
Device: 1 mA HD-tDCS — Participants will receive HD-tDCS at 1 mA for 30 minutes, for between 5-30 sessions.
  Arms: 1 mA Dosage Stimulation
Device: 2 mA HD-tDCS — Participants will receive HD-tDCS at 2 mA for 30 minutes, for between 5-30 sessions.
  Arms: 2 mA Dosage Stimulation
Device: 3 mA HD-tDCS — Participants will receive HD-tDCS at 3 mA for 30 minutes, for between 5-30 sessions.
  Arms: 3 mA Dosage Stimulation
Device: Sham — Participants will receive sham (placebo) HD-tDCS for 30 minutes, for between 5-30 sessions.
  Arms: Sham Stimulation

SUMMARY:
This study will test the effects of different doses of a form of non-invasive brain stimulation for the treatment of individuals with mild cognitive impairment (MCI) and dementia of the Alzheimer's Type (DAT).

DETAILED DESCRIPTION:
This research study is being done to learn important information about the effects of weak electrical stimulation on brain functioning in those with mild cognitive impairment (MCI) and dementia of the Alzheimer's type (DAT). The findings will help determine "how much" stimulation is needed to enhance memory and thinking abilities, how it affects brain functioning, and who is most likely to benefit. Ultimately, this information may guide treatment efforts for those at various stages of Alzheimer's disease. The study will use brain imaging to see whether these treatments change how participants learn and remember information. Functional magnetic resonance imaging (fMRI) and positron emission tomography (PET) scans will be used. The study will also use cognitive tests and questionnaires to examine whether participants' memory (and related abilities) change because of treatment. The study will enroll participants with a diagnosis of MCI or DAT. It is expected but not required that participants will be co-enrolled in the University of Michigan Memory and Aging Project (UM-MAP; HUM00000382).

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosis of Mild Cognitive Impairment (MCI) or dementia of the Alzheimer's type (DAT)
2. Must be MRI compatible, criteria that also apply for High Definition transcranial direct current stimulation (HD-tDCS; e.g., absence of metallic or electronic implants in the upper body or head)
3. Stable on relevant medications for at least 4 weeks prior to study enrollment

Exclusion Criteria:

1. Certain neurological diseases
2. Certain psychiatric conditions
3. Severe sensory impairment

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 269 (Actual)
Dates: Start 2019-04-01 (Actual); Primary Completion 2024-12-06 (Actual); Study Completion 2024-12-19 (Actual)

PRIMARY OUTCOMES:
Change in Lateral Temporal Cortex Connectivity | Baseline fMRI and post-intervention (after tDCS sessions 5 & 30)
  Graph Theory Analysis via fMRI using arbitrary units of connectivity strength

SECONDARY OUTCOMES:
Self-Report of Contentment with Memory | Baseline and post-intervention (after tDCS sessions 5 & 30)
  Multifactorial Memory Questionnaire (MMQ) Contentment Score
Self-Report of Memory Mistakes | Baseline and post-intervention (after tDCS sessions 5 & 30)
  Multifactorial Memory Questionnaire (MMQ) Ability Score
Self-Report of Memory Strategies Used | Baseline and post-intervention (after tDCS sessions 5 & 30)
  Multifactorial Memory Questionnaire (MMQ) Strategies Score
Change in Memory Functioning | Baseline and post-intervention (after tDCS sessions 5 & 30)
  Measured through change in the RBANS Delayed Memory Index
Change in Overall Fluid Cognitive Abilities | Baseline and post-intervention (after tDCS sessions 5 & 30)
  Measured through change in the NIH Toolbox Cognition Fluid Composite Score
Cumulative Working Memory Effects of HD-tDCS across daily sessions | Baseline Session through Session 6 then weekly up to final session
  Working memory accuracy measured by a discriminability ratio (2-back d' minus 0-back d') on a validated computerized N-Back task, measured after baseline (Session 1) and every intervention session (Sessions 2-6)
Cumulative Memory Accuracy Effects of HD-tDCS across daily sessions | Baseline Session through Session 6 then weekly up to final session
  Verbal memory accuracy measured by an accuracy score (percent correct) on a computerized Paired Associates task, measured after baseline (Session 1) and every intervention session (Sessions 2-6)
Cumulative Memory Reaction Time Effects of HD-tDCS across daily sessions | Baseline Session through Session 6 then weekly up to final session
  Verbal memory reaction time measured by a drift rate score (V; measured by the mean rate at which information is accumulated towards a boundary [correct or error response]) on a computerized Paired Associates task, measured after baseline (Session 1) and every intervention session (Sessions 2-6)
Tolerability of HD-tDCS | Prior to and immediately following each HD-tDCS session (<60 Minutes)
  Evaluated using standard questionnaires that arose from comprehensive reviews of the tDCS literature, this questionnaire was recently refined to include pre- and post-HD-tDCS symptom assessment. This will be administered prior to and immediately after every brain stimulation session (including sham).
Effectiveness of Blinding of HD-tDCS | Immediately following HD-tDCS sessions 5 and final session (<60 Minutes)
  Evaluated using a standard single question administered after every brain stimulation session (including sham).

OTHER OUTCOMES:
Change in Default Mode Network Connectivity | Baseline fMRI and post-intervention (after tDCS sessions 5 & 30)
  Graph Theory Analysis via fMRI using arbitrary units of connectivity strength to measure changes in the Default Mode Network, along with strength in and between other networks
Change in Inhibition Ability | Baseline and post-intervention (after tDCS sessions 5 & 30)
  A priori intent to measure through change in the NIH Toolbox Flanker Inhibitory Control and Attention Test Score
Change in Conceptualization Ability | Baseline and post-intervention (after tDCS sessions 5 & 30)
  A priori intent to measure through change in the NIH Toolbox Dimensional Change Card Sort Test Score
Change in Picture Sequence Memory | Baseline and post-intervention (after tDCS sessions 5 & 30)
  A priori intent to measure through change in the NIH Toolbox Picture Sequence Memory Test Score
Change in Working Memory Ability | Baseline and post-intervention (after tDCS sessions 5 & 30)
  A priori intent to measure through change in the NIH Toolbox List Sorting Working Memory Test Score
Change in Processing Speed | Baseline and post-intervention (after tDCS sessions 5 & 30)
  A priori intent to measure through change in the NIH Toolbox Pattern Comparison Processing Speed Test Score
Cumulative Working Memory Performance Effects of HD-tDCS across daily sessions | Baseline Session through Session 6 then weekly up to final session
  A priori intent to explore d' change for each N-Back task condition (2-back, 0-back) in order to understand the overall effect of the HD-tDCS on task performance.
Change in Global Cognition | Baseline and post-intervention (after tDCS sessions 5 & 30)
  Measured through change in the Total RBANS Score
Change in Visuospatial Functioning | Baseline and post-intervention (after tDCS sessions 5 & 30)
  Measured through change in the RBANS Visuospatial Index score
Change in Language Functioning | Baseline and post-intervention (after tDCS sessions 5 & 30)
  Measured through change in the RBANS Language Index score
Change in Attention | Baseline and post-intervention (after tDCS sessions 5 & 30)
  Measured through change in the RBANS Attention Index score
Change in Memory Functioning | Baseline and post-intervention (after tDCS sessions 5 & 30)
  Measured through change in the RBANS Immediate Memory Index score
Change in Cognitive Functioning | Baseline and post-intervention (after tDCS sessions 5 & 30)
  A priori intent to measure through changes in RBANS subtest scores
Cumulative Cognitive Change across Daily Consecutive Sessions | After each HD-tDCS Session, daily
  Measured through change in Cogstate or other comparable computerized cognitive testing scores across consecutive daily sessions

CONTACTS AND LOCATIONS:
Overall Officials: Benjamin Hampstead, PhD, Principal Investigator — Associate Professor
Locations (1):
- University of Michigan, Ann Arbor, Michigan, United States

IPD SHARING:
Plan to Share IPD: No